CLINICAL TRIAL: NCT02697019
Title: Internet-delivered Emotion Regulation Individual Therapy for Adolescents With NSSI - An Open Pilot Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Karolinska Institutet (Other)
Responsible Party: Principal Investigator, Clara Hellner Gumpert, PhD, Karolinska Institutet
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2015/1895-31/5
Record Dates: First submitted 2016-02-26; First posted 2016-03-02 (Estimated); Last update posted 2018-08-10 (Actual); Status verified 2018-08

CONDITIONS: Nonsuicidal Self-Injury
Keywords: Nonsuicidal Self-Injury (NSSI), Deliberate Self-Harm (DSH), Self-harm, Self-injury
MeSH Terms: conditions — Self-Injurious Behavior; Dyschromatosis symmetrica hereditaria 1

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Internet-delivered ERITA (Experimental)
  Interventions: Behavioral: Internet-delivered Emotion Regulation Individual Therapy for Adolescents

INTERVENTIONS:
Behavioral: Internet-delivered Emotion Regulation Individual Therapy for Adolescents

SUMMARY:
The primary aim is to investigate the effectiveness of an Internet-delivered Emotion Regulation Individual Therapy for Adolescents (ERITA) with nonsuicidal self-injury (NSSI).

ELIGIBILITY:
Inclusion Criteria:

A primary diagnosis of NSSI as defined in Section 3 in the fifth edition of the Diagnostic and Statistical Manual 5 of the American Psychiatric Association (DSM-5) < 1 NSSI episode during the past month At least one parent needs to commit to participate in the parent program

Exclusion Criteria:

Bipolar disorder I or primary psychosis Severe suicidal ideation Ongoing substance dependence Insertion/withdrawal of psychopharmacological substances within two months prior to the treatment Other acute primary axis I diagnosis (e.g. anorexia nervosa) that demand treatment in first hand Current life circumstances that would hinder the treatment (i.e. ongoing domestic abuse) insufficient Swedish language skills Cocurrent treatment with Mentalization based therapy (MBT) or Dialectical behavioral therapy (DBT)

Ages: 13 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 25 (Actual)
Dates: Start 2016-02 (Actual); Primary Completion 2017-12 (Actual); Study Completion 2017-12 (Actual)

PRIMARY OUTCOMES:
Deliberate Self-Harm Inventory - 9 item version | Baseline (30 days prior to treatment start), weekly (once a week following treatment start), post-treatment (12 weeks), and three and six months follow-up
  Change from baseline in self-harming behaviors when measures weekly, after 12 weeks, and at 3 and 6 months after treatment has ended

SECONDARY OUTCOMES:
Borderline Symptom List Behavior supplement (BSL-supplement) | Baseline (30 days prior to treatment start), weekly (once a week following treatment start), post-treatment (12 weeks), and three and six months follow-up
  Change from baseline in self-destructive behaviors when measures weekly, after 12 weeks, and at 3 and 6 months after treatment has ended
Difficulties in Emotion Regulation Scale -16 item version (DERS-16) | Baseline (30 days prior to treatment start), weekly (once a week following treatment start), post-treatment (12 weeks), and three and six months follow-up
  Change from baseline in difficulties in emotion regulation when measures weekly, after 12 weeks, and at 3 and 6 months after treatment has ended
Difficulties in Emotion Regulation Scale (DERS) | Baseline (7 days prior to treatment start), post-treatment (12 weeks), three and six months follow-up]
  Change from baseline in difficulties in emotion regulation after 12 weeks, at 3 and 6 months after treatment has ended
Borderline personality features in childhood (BPFS-C) | Baseline (7 days prior to treatment start), post-treatment (12 weeks), three and six months follow-up]
  Change from baseline in symptoms of borderline personality disorder after 12 weeks, at 3 and 6 months after treatment has ended
The Revised Child Anxiety and Depression Scale - Child and Parent rated (RCADS-C) | Baseline (7 days prior to treatment start), post-treatment (12 weeks), three and six months follow-up]
  Change from baseline in anxiety and depression after 12 weeks, at 3 and 6 months after treatment has ended
Suicidal Ideation Questionnaire (SIQ-JR) | Baseline (7 days prior to treatment start), post-treatment (12 weeks), three and six months follow-up]
  Change from baseline in suicidal ideation after 12 weeks, at 3 and 6 months after treatment has ended
Acceptance and Action Questionnaire (AAQ-7) | Baseline (7 days prior to treatment start), post-treatment (12 weeks), three and six months follow-up]
  Change from baseline in acceptance and action after 12 weeks, at 3 and 6 months after treatment has ended

OTHER OUTCOMES:
The treatment credibility scale | One week after treatment start
  Perceived treatment credibility
Working Alliance Inventory (WAI) short version | Three weeks after treatment start
  Perceived working alliance
The Client Satisfaction Questionnaire (CSQ) | Twelve weeks after treatment start
  Perceived client satisfaction
Adverse events | 12 weeks, and at 3 and 6 months after treatment has ended
  Adverse events
Adult ADHD Self-Report Scales (ASRS) | At baseline
  Self-reported symptoms of attention-deficit/hyperactivity disorder (ADHD)
Parental Psychological Flexibility (PPF) Questionnaire | Baseline (7 days prior to treatment start), post-treatment (12 weeks), three and six months follow-up]
  Change from baseline in parental psychological flexibility after 12 weeks, at 3 and 6 months after treatment has ended
The Coping with Children's Negative Emotions Scale Adolescent Version (CCNES-A) | Baseline (7 days prior to treatment start), post-treatment (12 weeks), three and six months follow-up]
  Change from baseline in parental coping after 12 weeks, at 3 and 6 months after treatment has ended
The Parenting Sense of Competence (PSOC) Scale | Baseline (7 days prior to treatment start), post-treatment (12 weeks), three and six months follow-up]
  Change from baseline in parental coping after 12 weeks, at 3 and 6 months after treatment has ended

CONTACTS AND LOCATIONS:
Locations (1):
- Karolinska Institutet, Stockholm, Sweden

REFERENCES:
- [Derived] Bjureberg J, Sahlin H, Hedman-Lagerlof E, Gratz KL, Tull MT, Jokinen J, Hellner C, Ljotsson B. Extending research on Emotion Regulation Individual Therapy for Adolescents (ERITA) with nonsuicidal self-injury disorder: open pilot trial and mediation analysis of a novel online version. BMC Psychiatry. 2018 Oct 11;18(1):326. doi: 10.1186/s12888-018-1885-6. PMID 30305103